CLINICAL TRIAL: NCT03186716
Title: Effects of Colostrum Supplement on Intestinal Permeability in Hospitalized Patients With Enteral Feeding in Intensive Care Unit
Brief Title: A Trial of Enteral Colostrum on Intestinal Permeability in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Ghazaleh Eslamian, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017670
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness
Keywords: Colostrum; Enteral Nutrition; Intestinal Permeability; Intensive Care Unit
MeSH Terms: conditions — Critical Illness | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colostrum (Experimental): Intervention patients will be received enteral formula and colostrum powder 20 g/kg/day given via nasogastric tube as boluses q 4hrs.
  Interventions: Dietary Supplement: Colostrum
- Maltodextrin (Placebo Comparator): Control patients will be received enteral formula and maltodextrin mixed in with water and given via nasogastric tube as boluses q 4hrs.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Colostrum — Enteral colostrum 20g/day powdered colostrum to be mixed in with water and given via nasogastric tube q4 hrs.
  Other Names: Bovine Colostrum
  Arms: Colostrum
Dietary Supplement: Maltodextrin — Control patients will be received enteral formula and maltodextrin mixed in with water and given via nasogastric tube as boluses q 4hrs.
  Arms: Maltodextrin

SUMMARY:
The effects of colostrum on intestinal permeability in critical ill patients has not been investigated. In current trial, intensive care unit patients with enteral feeding will receive either enteral colostrum or maltodextrin as placebo.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in general intensive care unit (ICU) in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. Intervention patients will be received 20 g/day of colostrum along with enteral formula and control patients will be received maltodextrin along with enteral formula. Patients will be evaluated for plasma endotoxin and plasma zonulin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) admitted to ICU
* Start of study intervention within 48 hours after ICU admission
* Expected to require enteral nutrition for at least 72 hours aiming for full enteral nutrition and receive at least 80 percent of enteral formula during the first 48 hour
* Written informed consent of patient or written informed consent of legal representative

Exclusion Criteria:

* Enrollment in a related ICU interventional study
* Requiring other specific enteral nutrition for medical reason
* Death or Discharge before 5th day
* Having any contra-indication to receive enteral nutrition
* Pregnant patients or lactating with the intent to breastfeed
* BMI <18 or > 40.0 kg/m2
* Have life expectancy of <6 mo
* Patients who are moribund
* History of allergy or intolerance to the study product components
* Receiving colostrum during two weeks before start study product
* Have other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-11 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline plasma endotoxin concentration at 10 days | baseline, Day 5, Day 10
  The levels of plasma endotoxin
Change from Baseline plasma zonulin concentration at 10 days | baseline, Day 5, Day 10
  The levels of plasma zonulin

SECONDARY OUTCOMES:
Gastrointestinal complications | Day 10
  abdominal distention, vomiting, diarrhea and constipation
Mortality in ICU | Day 10
  Mortality rate
length of stay in ICU | Day 10
  Duration of stay in ICU
incidence of severe sepsis | Day 10
  according to the American College of Chest Physicians and the Society of Critical Care Medicine

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Eslamian, MS,PhDcandid, Principal Investigator — National Nutrition and Food Technology Research Institute Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JW, Jeon WK, Kim EJ. Combined effects of bovine colostrum and glutamine in diclofenac-induced bacterial translocation in rat. Clin Nutr. 2005 Oct;24(5):785-93. doi: 10.1016/j.clnu.2005.04.004. PMID 15919136
- [Background] Rathe M, Muller K, Sangild PT, Husby S. Clinical applications of bovine colostrum therapy: a systematic review. Nutr Rev. 2014 Apr;72(4):237-54. doi: 10.1111/nure.12089. Epub 2014 Feb 26. PMID 24571383
- [Background] Benson KF, Carter SG, Patterson KM, Patel D, Jensen GS. A novel extract from bovine colostrum whey supports anti-bacterial and anti-viral innate immune functions in vitro and in vivo: I. Enhanced immune activity in vitro translates to improved microbial clearance in animal infection models. Prev Med. 2012 May;54 Suppl:S116-23. doi: 10.1016/j.ypmed.2011.12.023. Epub 2011 Dec 28. PMID 22227281
- [Background] Halasa M, Maciejewska D, Baskiewicz-Halasa M, Machalinski B, Safranow K, Stachowska E. Oral Supplementation with Bovine Colostrum Decreases Intestinal Permeability and Stool Concentrations of Zonulin in Athletes. Nutrients. 2017 Apr 8;9(4):370. doi: 10.3390/nu9040370. PMID 28397754
- [Background] Yoon JY, Park SJ, Cheon JH. Effect of Colostrum on the Symptoms and Mucosal Permeability in Patients with Irritable Bowel Syndrome: A Randomized Placebo-controlled Study. Intest Res. 2014 Jan;12(1):80-2. doi: 10.5217/ir.2014.12.1.80. Epub 2014 Jan 28. No abstract available. PMID 25349570
- [Derived] Eslamian G, Ardehali SH, Baghestani AR, Vahdat Shariatpanahi Z. Effects of early enteral bovine colostrum supplementation on intestinal permeability in critically ill patients: A randomized, double-blind, placebo-controlled study. Nutrition. 2019 Apr;60:106-111. doi: 10.1016/j.nut.2018.10.013. Epub 2018 Oct 12. PMID 30551120